CLINICAL TRIAL: NCT02610062
Title: A Phase 1 Study Evaluating Safety, Tolerability, and Pharmacokinetics of Escalating Doses of AGS67E Given as Monotherapy in Subjects With Acute Myeloid Leukemia (AML)
Brief Title: A Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Escalating Doses of AGS67E Given as Monotherapy in Subjects With Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision by sponsor
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS67E-15-2
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — AGS67E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AGS67E 1.2 mg/kg Schedule 1 (Experimental): Participants will receive 1.2 mg/kg of AGS67E as an intravenous infusion once every three weeks (Q3).
  Interventions: Drug: AGS67E
- AGS67E 1.8 mg/kg Schedule 1 (Experimental): Participants will receive 1.8 mg/kg of AGS67E as an intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- AGS67E 2.4 mg/kg Schedule 1 (Experimental): Participants will receive 2.4 mg/kg of AGS67E as an intravenous infusion once every three weeks.
  Interventions: Drug: AGS67E
- AGS67E 0.6 mg/kg Schedule 2 (Experimental): Participants will receive 0.6 mg/kg of AGS67E once weekly for three weeks.
  Interventions: Drug: AGS67E
- AGS67E 0.9 mg/kg Schedule 2 (Experimental): Participants will receive 0.9 mg/kg of AGS67E once weekly for three weeks.
  Interventions: Drug: AGS67E

INTERVENTIONS:
Drug: AGS67E — Intravenous (IV) infusion

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of AGS67E in subjects with acute myeloid leukemia (AML) and determine a safe dose for future development. In addition, this study will assess the pharmacokinetics (PK), the immunogenicity, and the anti-leukemic activity of AGS67E.

DETAILED DESCRIPTION:
The study will sequentially evaluate AGS67E given as a 30 minute intravenous (IV) infusion in two different schedules: once every 3 weeks (Q3) and then once weekly for 3 weeks.

The dose escalation follows a 3 + 3 design.

The Data Review Team may expand any dose level or intermediate dose level that has been deemed safe and resulted in at least one subject with a Composite Complete Remission (CRc). An expansion cohort may enroll up to 15 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has morphologically documented primary or secondary AML by the World Health Organization (WHO) criteria (2008) and fulfills one of the following:

  * Refractory to at least 1 cycle of induction chemotherapy
  * Relapsed after achieving remission with a prior therapy
  * Patients with untreated AML who are either unwilling or unable to undergo high-dose induction/consolidation intensive chemotherapy
* Circulating blasts < 20,000 (cytoreduction with hydroxyurea is allowed)
* Eastern Cooperative Oncology Group performance score (ECOG) ≤ 2
* Subject has adequate renal function: serum creatinine ≤ 2.0 mg/dL and estimated creatinine clearance of ≥ 30 mL/min by the Cockcroft-Gault equation
* Subject has a total bilirubin ≤ 1.5 x upper limit of normal (ULN), albumin ≥ 2.5 g/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Negative pregnancy test in women of child bearing potential
* Sexually active fertile subjects, and their partners, must agree to use medically accepted double-barrier methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the study and at least 6 weeks after termination of study therapy

Exclusion Criteria:

* Subject has a diagnosis of acute promyelocytic leukemia
* Subject has preexisting sensory or motor neuropathy Grade ≥ 2 at baseline
* Subject has received small molecule therapy, radiotherapy, immunotherapy, monoclonal antibodies, investigational drug, or chemotherapy within 14 days before first dose of study drug, with the exception of hydroxyurea
* P-gp inducers/inhibitors or strong CYP3A inhibitors within 14 days before the first dose of drug, with the exception of the antibiotics/ antifungals used as prophylaxis and/or supportive care
* Any Grade ≥ 2 persistent non-hematological toxicity related to allotransplant
* Graft-Versus-Host Disease (GVHD) therapy within 6 weeks before the first dose of study drug; low dose steroids (≤ 10mg) allowed
* Subject has known current central nervous system (CNS) disease
* Active angina or Class III or IV Congestive Heart Failure (New York Heart Association CHF Functional Classification System) or clinically significant cardiac disease within 6 months of the first dose of study drug, including myocardial infarction, unstable angina, Grade 2 or greater peripheral vascular disease, congestive heart failure, uncontrolled hypertension, or arrhythmias not controlled by medication
* Subject has clinical evidence of Disseminated Intravascular Coagulation (DIC)
* Subject has known positivity for human immunodeficiency virus (HIV)
* Subject has know positivity for Hepatitis B surface antigen test or Hepatitis C Antibody
* Subject has an uncontrolled active infection requiring treatment and fever 38.3°C or higher 48 hours before the first dose of study drug. Controlled infections (i.e. 3 negative cultures completing antibiotics and/or stable fungal infection in therapy are allowed provided the subject has a temperature of <38.3°C within 48 hours of the first dose of study drug
* Subject has known sensitivity to any of the components of the investigational product AGS67E:

  * AGS67E
  * L-Histidine
  * α-trehalose dihydrate or
  * polysorbate 20
* Major surgery within 28 days of the first dose of study drug
* Subject is pregnant or lactating
* Subject has a condition or situation which may put the subject at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of adverse events | Up to 24 months

SECONDARY OUTCOMES:
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose escalation part: Concentration at the end of infusion (CEOI) | Escalation Q3 weeks dosing: up to Day 15 for Cycle 1, Day 8 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Escalation weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose expansion part: Concentration at the end of infusion (CEOI) | Expansion Q3 weeks dosing: up to Day 8 for Cycle 1, Day 3 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Expansion weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose escalation part: Maximum observed concentration (Cmax) | Escalation Q3 weeks dosing: up to Day 15 for Cycle 1, Day 8 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Escalation weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose expansion part: Maximum observed concentration (Cmax) | Expansion Q3 weeks dosing: up to Day 8 for Cycle 1, Day 3 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Expansion weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for Monomethyl Auristatin E (MMAE) in dose escalation part: Time to maximum concentration (Tmax) | Escalation Q3 weeks dosing: up to Day 15 for Cycle 1, Day 8 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Escalation weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for Monomethyl Auristatin E (MMAE) in dose expansion part: Time to maximum concentration (Tmax) | Expansion Q3 weeks dosing: up to Day 8 for Cycle 1, Day 3 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Expansion weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose escalation part: Partial area under the serum concentration-time curve (AUC) | Escalation Q3 weeks dosing: up to Day 15 for Cycle 1, Day 8 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Escalation weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose expansion part: Partial area under the serum concentration-time curve (AUC) | Expansion Q3 weeks dosing: up to Day 8 for Cycle 1, Day 3 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Expansion weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose escalation part: Terminal or apparent terminal half-life (t1/2) | Escalation Q3 weeks dosing: up to Day 15 for Cycle 1, Day 8 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Escalation weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose expansion part: Terminal or apparent terminal half-life (t1/2) | Expansion Q3 weeks dosing: up to Day 8 for Cycle 1, Day 3 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Expansion weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose escalation part: Systemic clearance (CL) | Escalation Q3 weeks dosing: up to Day 15 for Cycle 1, Day 8 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Escalation weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose expansion part: Systemic clearance (CL) | Expansion Q3 weeks dosing: up to Day 8 for Cycle 1, Day 3 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Expansion weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose escalation part: Volume of distribution at steady state (Vss) | Escalation Q3 weeks dosing: up to Day 15 for Cycle 1, Day 8 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Escalation weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Pharmacokinetic parameter for total antibody (TAb), antibody drug conjugate (ADC), and Monomethyl Auristatin E (MMAE) in dose expansion part: Volume of distribution at steady state (Vss) | Expansion Q3 weeks dosing: up to Day 8 for Cycle 1, Day 3 for Cycle 2, predose in subsequent cycles up to an average of 12 months. Expansion weekly dosing: up to Day 22 for Cycles 1, 2 and predose in subsequent cycles up to an average of 12 months
Incidence of Anti-Drug Antibody (ADA) formation to the fully human monoclonal antibody (AGS67C) and antibody-drug conjugate (AGS67E) | Up to 24 months
Complete remission (CR) rate | Up to 24 months
Composite CR (CRc) rate | Up to 24 months
Best overall response rate | Up to 24 months
  Best overall response rate is defined as the percentage of subjects who experience a best overall response of CRc, partial response (PR) or morphologic leukemia-free state (MLFS)
Duration of remission | Up to 24 months
  Duration of remission is the duration of CRc, CR, completion remission with incomplete hematologic recovery (CRi) and completion remission with incomplete platelet recovery (CRp)
Duration of response | Up to 24 months
  Duration of response is CRc, PR and MLFS

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (4):
- United States (3):
  - Site US0006, Duarte, California
  - Site US0004, New York, New York
  - Site US0001, Houston, Texas
- Site CA0010, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on ACSR website — https://astellasclinicalstudyresults.com/study.aspx?ID=340